CLINICAL TRIAL: NCT03009435
Title: RMOS Study : Impact of Manual Rotation of Occiput Posterior Position on Operative Delivery Rate
Brief Title: RMOS Study : Impact of Manual Rotation of Occiput Posterior Position on Operative Delivery Rate (RMOS)
Acronym: RMOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-A01456-45
Record Dates: First submitted 2016-12-19; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Fetal Manual Rotation

ARMS (2):
- prophylactic manual rotation (Experimental): Only obstetricians will participate in the study. Manual rotation is performed at full dilatation.The technique employed will be at the discretion of the operator performing the procedure :
  * Tarnier and Chantreuil technique
  * or SOGC technique
  Interventions: Other: prophylactic manual rotation
- expectative management (No Intervention): Expectative management . No manual rotation

INTERVENTIONS:
Other: prophylactic manual rotation
  Arms: prophylactic manual rotation

SUMMARY:
Introduction:

The frequency of fetuses in occiput posterior position during labor is approximately 20 %, in which 5% remain occiput posterior at the end of labor. Occiput posterior position is associated with higher risks of caesarean deliveries and operative vaginal deliveries. The manual rotation to promote rotation from a posterior to an anterior position has been proposed to reduce the extraction rate. There is no randomised trial comparing the effect of manual rotation and expectant management. We propose a protocol for a prospective, monocentric, randomised controlled clinical trial in order to show that the rate of spontaneous vaginal delivery is higher with manual rotation of occiput posterior position than with an expectative management.

Methods:

Every 37 weeks with a singleton pregnancy with a clinical occiput posterior position suspicion confirmed by a transabdominal ultrasound at full dilatation will be eligible. Participants will be randomised to either prophylactic manual rotation (experimental group) or expectative management (control group). Based on an alpha value of 0.05 and gaining 20% for spontaneous vaginal delivery, 238 participants will need to be enrolled.

The primary outcome will be spontaneous vaginal delivery. Secondary outcomes will be operative delivery rate (caesarean section , vacuum or forceps deliveries), significant maternal and perinatal mortality/morbidity.

Analysis will be by intention-to-treat averaging a 24-month period.

ELIGIBILITY:
1. Inclusion Criteria:

   * age ≥ 18 years
   * singleton pregnancy

     -≥37 weeks of gestation
   * planned vaginal birth
   * cephalic presentation
   * occiput posterior position confirmed by ultrasound at full dilatation
2. Exclusion Criteria:

   * withdrawal of consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of spontaneous vaginal delivery | At the time of delivery

REFERENCES:
- [Derived] Verhaeghe C, Corroenne R, Spiers A, Descamps P, Gascoin G, Bouet PE, Parot-Schinkel E, Legendre G. Delivery Mode After Manual Rotation of Occiput Posterior Fetal Positions: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):999-1006. doi: 10.1097/AOG.0000000000004386. PMID 33957650
- [Derived] Verhaeghe C, Parot-Schinkel E, Bouet PE, Madzou S, Biquard F, Gillard P, Descamps P, Legendre G. The impact of manual rotation of the occiput posterior position on spontaneous vaginal delivery rate: study protocol for a randomized clinical trial (RMOS). Trials. 2018 Feb 14;19(1):109. doi: 10.1186/s13063-018-2497-7. PMID 29444695